CLINICAL TRIAL: NCT03805802
Title: Influence of a Liquid Oat Bran Product on Blood Glucose in Patients With Poorly Controlled Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stoffwechselzentrum Rhein - Pfalz (Other)
Collaborators: Glucanova AB (Unknown)
Responsible Party: Principal Investigator, Dr. Per Humpert, Director of Stoffwechselzentrum Rhein - Pfalz, Stoffwechselzentrum Rhein - Pfalz
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 012019
Record Dates: First submitted 2019-01-13; First posted 2019-01-16 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus, Type 2; Obesity; Overweight; Metabolic Syndrome
Keywords: fiber; type 2 diabetes; dietary intervention; weight loss; glucose control; obesity; overweight; metabolic syndrome; oats
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Overweight; Metabolic Syndrome; Weight Loss

STUDY DESIGN:
Intervention Model Description: First 6 weeks double blinded vs. a reference product and second 6 weeks open label both groups receive the test product in the second 6 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigator receives reference product and the test product in boxes labelled "stratus" "nimbus" and "cumulus". first 6 weeks participants are randomly assigned to "stratus" or "nimbus" and the second 6 weeks participants all receive "cumulus".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active product (Experimental): Once daily ad libitum consumption of one package of the fiber product 6 weeks (blinded phase). Once daily ad libitum consumption of one package of the fiber product 6 weeks (open phase).
  Interventions: Other: active product
- reference product (Placebo Comparator): Once daily ad libitum consumption of one package of placebo during 6 weeks (blinded phase). Once daily ad libitum consumption of one package of the fiber product 6 weeks (open phase).
  Interventions: Other: active product; Other: reference product

INTERVENTIONS:
Other: active product — Once daily consumption over the period of the study
  Other Names: LOB; Liquid Oat Bran; High fiber product
Other: reference product — Once daily consumption over the period of the study
  Other Names: placebo food product
  Arms: reference product

SUMMARY:
This study evaluates the effects of an ad libitum addition of a high fiber product to the regular diet of type 2 diabetes patients on body weight and blood sugar control. In the first 6 weeks half of the participants will receive the high fiber test product and half a reference product without fiber. After the first 6 weeks both groups will be switched to the high fiber product.

DETAILED DESCRIPTION:
It has previously been shown that an increase in the consumption of fiber improves glucose control in type 2 diabetes. In addition, previous pilot studies have shown that a diet solely based on oat flakes can improve insulin sensitivity and glucose control in poorly controlled type 2 diabetes. Recent clinical data indicates, that early hyperglycemia can be normalized by a diet high in fiber. In this controlled pilot study, a food containing liquid oat bran high in fiber will be studied in type 2 diabetes patients with inadequate glucose control that are treated with oral medication or with additional once-daily insulin only against a reference product. 30 patients will be treated with the oat bran product or reference product over a period of 6 weeks in a double blinded approach, hereafter all participants will be switched to the oat bran product. The primary endpoint will be fasting glucose after 6 weeks. Secondary endpoints will be long-term glucose control as measured by HbA1c, self-documented glucose as well as the body weight and body mass index.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes with inadequate glucose control and a HbA1c >7,5 and < 9%
* Treatment with all oral antidiabetic medication or injectable GLP-1 analogues
* BMI 28,0-39,9 kg/m²
* Age 30-70 years

Exclusion Criteria:

* insulin treatment
* Psychiatric Disease
* Acute Infections
* Alcohol or drug abuse
* Acute diverticulitis
* Malignant tumors or hematologic disorders
* Heart failure NYHA III-IV
* Acute coronary syndrome
* Chronic kidney disease > Stage 3 (KDOQI)
* Pregnancy or Lactation
* Previous bariatric interventions

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Fasting glucose | 6 weeks
  Change in the concentratino of fasting venous glucose of daily LOB consumption in mg/dl as compared to the change in fasting glucose for the placebo group at 6 weeks.

SECONDARY OUTCOMES:
Fasting glucose | 12 weeks
  Change in the concentratino of fasting venous glucose of daily LOB consumption in mg/dl as compared to the change in fasting glucose for the placebo group at 12 weeks.
HBA1c | 6 weeks
  long-term glucose control as measured by the concentratino of HbA1c concentration in %
HBA1c | 12 weeks
  long-term glucose control as measured by the concentratino of HbA1c concentration in %
Self-documented glucose | 6 weeks
  Self-monitored glucose levels extracted from glucometers as a mean of the previous two weeks before study visits in mg/dl
Self-documented glucose | 12 weeks
  Self-monitored glucose levels extracted from glucometers as a mean of the previous two weeks before study visits in mg/dl
Weight | 6 weeks
  Chenge in body Weight in kg
Weight | 12 weeks
  Chenge in body Weight in kg
BMI | 6 weeks
  Body Mass Index
BMI | 12 weeks
  Body Mass Index
Lipid metabolism: Serum triglycerides | 6 weeks
  Markers of lipid metabolism at 6 weeks: triglycerides (mg/dl)
Lipid metabolism: Serum triglycerides | 12 weeks
  Markers of lipid metabolism at 12 weeks: triglycerides (mg/dl)
Lipid metabolism: apolipoprotein A (mg/dl) | 6 weeks
  Markers of lipid metabolism at 6 weeks: apolipoprotein A (mg/dl)
Lipid metabolism: apolipoprotein A (mg/dl) | 12 weeks
  Markers of lipid metabolism at 12 weeks: apolipoprotein A (mg/dl)
Lipid metabolism: Apolipoprotein B mg/dl | 6 weeks
  Markers of lipid metabolism at 6 weeks: Apolipoprotein B mg/dl
Lipid metabolism: Apolipoprotein B mg/dl | 12 weeks
  Markers of lipid metabolism at 12 weeks: Apolipoprotein B mg/dl
Lipid metabolism: Apolipoprotein B / Apolipoprotein A ratio | 6 weeks
  Metabolism at 6 weeks: Apolipoprotein B mg/dl / Apolipoprotein A mg/dl ratio
Lipid metabolism: Apolipoprotein B / Apolipoprotein A ratio | 12 weeks
  Markers of lipid metabolism at 12 weeks: Apolipoprotein B mg/dl / Apolipoprotein A mg/dl ratio
Lipid metabolism: HDL-cholesterol | 6 weeks
  Markers of lipid metabolism at 6 weeks: HDL-cholesterol mg/dl
Lipid metabolism: HDL-cholesterol | 12 weeks
  Markers of lipid metabolism at 12 weeks: HDL-cholesterol mg/dl
Lipid metabolism: LDL- cholesterol mg/dl | 6 weeks
  Markers of lipid metabolism at 6 weeks: LDL- cholesterol mg/dl
Lipid metabolism: LDL- cholesterol mg/dl | 12 weeks
  Markers of lipid metabolism at 12 weeks: LDL- cholesterol mg/dl
Microbiome | 6 weeks
  Microbiome in faeces samples at 6 weeks
Microbiome | 12 weeks
  Microbiome in faeces samples at 12 weeks
Inflammation: Il-6 | 6 weeks
  Markers of inflammation at 6 weeks IL-6 in ng/ml
Inflammation: hsCRP | 6 weeks
  Markers of inflammation at 6 weeks hsCRP mg/l
Inflammation: Il-6 | 12 weeks
  Markers of inflammation at 12 weeks IL-6 in ng/ml
Inflammation: hsCRP | 12 weeks
  Markers of inflammation at 12 weeks hsCRP mg/l

OTHER OUTCOMES:
Systolic lood pressure | 6 weeks
  Systolic blood pressure left arm 6 weeks in mm/Hg
Diastolic blood pressure | 6 weeks
  Diastolic blood pressure left arm 6 weeks in mm/Hg
Systolic blood pressure | 12 weeks
  Systolic blood pressure left arm 12 weeks in mm/Hg
Diastolic blood pressure | 12 weeks
  Diastolic blood pressure left arm 12 weeks in mm/Hg
Waist circumference | 6 weeks
  Waist circumference at 6 weeks in cm
Waist circumference | 12 weeks
  Waist circumference at 12 weeks in cm

CONTACTS AND LOCATIONS:
Overall Officials: Per M Humpert, M. D., Principal Investigator — Director of Stoffwechselzentrum Rhein-Pfalz
Locations (1):
- Stoffwechselzentrum Rhein-Pfalz, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No